CLINICAL TRIAL: NCT06976840
Title: Rapid Antidepressant Dynamics in Acute Neuromodulation Treatments
Acronym: RADIANT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marta Peciña, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Marta Peciña, MD PhD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: STUDY24040131
Record Dates: First submitted 2025-04-30; First posted 2025-05-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Depression; Major Depressive Disorder
Keywords: theta burst stimulation; reinforcement learning; neuroimaging
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: This is a mechanistic trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Salience Network Target (Other): Intermittent/Sham/Continuous TBS, counterbalanced in order.
  Interventions: Device: Intermittent theta burst stimulation; Device: Sham theta burst stimulation; Device: Continuous theta burst stimulation
- Default Mode Network Target (Experimental): Intermittent/Sham/Continuous TBS, counterbalanced in order.
  Interventions: Device: Intermittent theta burst stimulation; Device: Sham theta burst stimulation; Device: Continuous theta burst stimulation

INTERVENTIONS:
Device: Intermittent theta burst stimulation — Aimed at potentiating the stimulation target.
Device: Sham theta burst stimulation — No effect is expected on stimulation target
Device: Continuous theta burst stimulation — Aimed at depotentiating the stimulation target

SUMMARY:
The goal of this clinical trial is to learn how different types of non-invasive brain stimulation affect mood and brain function in adults with major depressive disorder (MDD). It will also study how brain stimulation may work together with antidepressant treatments.

The main questions this study aims to answer are:

How do different patterns of brain stimulation affect mood in people with depression?

Do brain networks involved in emotion and self-reflection respond differently depending on the type of stimulation?

What are the combined effects of brain stimulation and antidepressant treatments on mood and brain activity?

Researchers will compare different brain stimulation patterns and target areas to understand their individual and combined effects.

Participants will:

Receive three types of brain stimulation (intermittent, continuous, and sham) in different sessions

Undergo MRI scans during the administration of either a fast-acting or conventional antidepressant

Complete mood assessments during the scan and for one week after each session

This study may help identify brain-based strategies to improve treatment for depression.

DETAILED DESCRIPTION:
This mechanistic clinical trial will investigate the role of large-scale brain networks in modulating mood responses in adults with major depressive disorder (MDD) using non-invasive neuromodulation and neuroimaging. The study will focus on the salience network (SN), default mode network (DMN), and functional connectivity (FC) between them, given prior evidence linking these systems to mood regulation and antidepressant response.

Using a 2x3 factorial design, 200 participants with MDD will be randomized to receive theta burst stimulation (TBS) targeting either the SN or the DMN (between-subject factor). Each participant will complete three within-subject TBS sessions one week apart: intermittent TBS (iTBS), continuous TBS (cTBS), and sham stimulation. TBS will be delivered over individualized fMRI-based targets derived from prior resting-state connectivity maps.

Following each stimulation session, participants will complete an MRI protocol that includes administration of either a fast-acting or conventional antidepressant, as well as resting-state functional imaging.

Primary neural outcomes include changes in activation and connectivity within and between SN and DMN regions, measured using task-based and resting-state fMRI. Behavioral outcomes include mood ratings acquired repeatedly during the scanning session and via daily remote assessments for one week post-stimulation.

This design allows for within-subject comparison of the acute and sub-acute effects of different TBS patterns, and between-subject comparison of SN- vs. DMN-targeted stimulation. The study aims to identify brain circuits that can be engaged or modulated to enhance treatment response in depression, with the longer-term goal of informing precision neuromodulation strategies.

Note: Certain information is withheld to protect the scientific integrity of the study design.

ELIGIBILITY:
Inclusion criteria:

1. Adults ages 18-55 (~60% female).
2. Diagnosis of Major Depressive Disorder (MDD) with or without comorbid anxiety disorders (e.g., panic disorder) or Axis II disorders.
3. Psychotropic-free at enrollment.

Exclusion Criteria:

1. being pregnant or breastfeeding;
2. diagnosis of psychotic depression, schizophrenia, bipolar disorder, or other Axis I disorders, except for anxiety disorders;
3. severe substance use (excluding nicotine) in the last 2 months as determined by using the MINI, a structured interview that uses the Diagnostic and Statistical Manual of Mental Disorders;
4. requiring immediate hospitalization;
5. epilepsy or conditions requiring an anticonvulsant;
6. receiving vagus nerve stimulation, electroconvulsive therapy (ECT), or TMS in the last 2 months;
7. currently taking or have taken within the last 21 days psychiatric medication or augmenting agents;
8. receiving depression-specific psychotherapy;
9. actively suicidal or considered a high suicide risk;
10. enrolled in another study; or
11. MRI/TMS contraindication as determined by the fMRI and TMS screening questionnaires

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2030-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Bold Signal Change in the Salience Network During the fMRI Experiment | Assessed at approximately day 7, day 14, and day 21 following baseline.
  Change in blood oxygenation level-dependent (BOLD) signal within the salience network (SN), measured during the fMRI experiment. Comparisons is made across transcranial magnetic stimulation conditions: intermittent theta burst stimulation (iTBS) vs. sham TBS (sTBS), and continuous TBS (cTBS) vs. sTBS. SN activation is assessed using fMRI contrasts sensitive to expectancy-induced neural modulation.
BOLD Signal Change in the Default Mode Network During the fMRI Experiment | Assessed at approximately day 7, day 14, and day 21 following baseline.
  Change in blood oxygenation level-dependent (BOLD) signal within the default mode network (DMN), measured during the fMRI experiment. Comparisons is made across transcranial magnetic stimulation conditions: intermittent theta burst stimulation (iTBS) vs. sham TBS (sTBS), and continuous TBS (cTBS) vs. sTBS. DMN activation is assessed using fMRI contrasts sensitive to expectancy-induced neural modulation.
Changes in Mood Ratings Following TBS and the fMRI Experiment | Baseline
  Change in self-reported mood, coded as a binary indicator of perceived mood improvement (yes/no), is assessed after each TBS session (iTBS, cTBS, sTBS) during the fMRI task. Participants are considered to show mood improvement if their post-stimulation average mood rating across trials increased relative to baseline. Between-condition comparisons (iTBS vs. sTBS; cTBS vs. sTBS) are conducted to evaluate the acute effects of TBS on mood reactivity.
Subcute Mood Change Following TBS and the fMRI experiment | Approximately at day 7, 14, and 21
  Change in depressive symptoms is assessed using the 16-item Quick Inventory of Depressive Symptomatology - Self-Report (QIDS-SR16; range: 0-27), where higher scores indicate greater depressive symptom severity. The QIDS-SR16 evaluates core domains of depression, including mood, interest, sleep, appetite, and concentration, over the past 7 days. Between-session changes (baseline to days 7, 14, and 21) are analyzed to assess subacute mood effects of intermittent TBS (iTBS), continuous TBS (cTBS), and sham TBS (sTBS) and the fMRI experimental manipulation.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Pecina, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Bellefield Towers, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Sharing plans will be defined after funding.